CLINICAL TRIAL: NCT03783039
Title: A Prospective, RCT Evaluating the Safety and Hemostatic Effectiveness of SURGICEL Powder in Controlling Mild or Moderate Parenchymal or Soft Tissue Intraoperative Bleeding During Surgery in Chinese Adult Subjects
Brief Title: The SURGICEL® Powder Mild or Moderate Parenchymal or Soft Tissue Intraoperative Bleeding (China Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOS_2017_02
Record Dates: First submitted 2018-12-06; First posted 2018-12-20 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Hemorrhage
Keywords: bleeding; broad area oozing bleeding; hemostat; topical hemostatic agents; adjunctive hemostats
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SURGICEL Powder (Experimental): SURGICEL Powder is an absorbable hemostat that is oxidized regenerated cellulose in a powder form
  Interventions: Device: SURGICEL Powder
- SURGICEL Original (Active Comparator): SURGICEL Original is an bsorbable hemostat that is oxidized regenerated cellulose in a fabric form
  Interventions: Device: SURGICEL Original

INTERVENTIONS:
Device: SURGICEL Powder — Surgeon to perform surgical procedure according to standard of care. If randomized to SURGICEL Powder, the product will be be applied to the first appropriate TBS with mild or moderate bleeding in parenchyma or soft tissue where conventional methods of control (i.e. suture, ligature, cautery) are ineffective or impractical.
  Arms: SURGICEL Powder
Device: SURGICEL Original — Surgeon to perform surgical procedure according to standard of care. If randomized to SURGICEL Original, the product will be be applied to the first appropriate TBS with mild or moderate bleeding in parenchyma or soft tissue where conventional methods of control (i.e. suture, ligature, cautery) are ineffective or impractical.
  Arms: SURGICEL Original

SUMMARY:
This is a single blind, randomized, prospective study comparing SURGICEL Powder with SURGICEL Original (control arm) as an adjunct to achieve hemostasis in the control of capillary, venous, and small arterial hemorrhage when ligation or other conventional methods of control are impractical or ineffective during surgery (open, laparoscopic, or thoracoscopic) in Chinese adult subjects.

DETAILED DESCRIPTION:
This is a single blind, randomized, prospective study comparing SURGICEL Powder with SURGICEL Original (control arm) as an adjunct to achieve hemostasis in the control of capillary, venous, and small arterial hemorrhage when ligation or other conventional methods of control are impractical or ineffective during surgery (open, laparoscopic, or thoracoscopic) in Chinese adult subjects.

After application of either SURGICEL Powder or SURGICEL Original, the target bleeding site (TBS) will be assessed for hemostasis (no detectable bleeding) at 3, 5, and 10 minutes from application and prior to initiation of final fascial closure on open surgery or port site closure in laparoscopic or thoracoscopic procedures.

All enrolled subjects will be observed post-operatively through discharge and followed up at 30 days (+14 days) and at 6 months (+/-30 days) post-surgery via phone call or office visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged ≥18 years requiring elective/non-emergent open or laparoscopic general, gynecological, or cardiothoracic surgical procedures.
2. Subject or authorized representative has signed the approved Informed Consent.
3. Subject(s) whose platelet count is ≥100,000 per microliter and International Normalized Ratio (INR) is <1.5 prior to 24 hours of surgery.
4. Presence of an appropriate TBS identified intra-operatively by the surgeon.
5. Subject(s) undergoing cardiothoracic surgery with anticoagulation must have anticoagulation reversed prior to TBS identification and treatment.

Exclusion Criteria:

1. Female subjects who are pregnant or nursing.
2. Subject on heparin within 12 hours prior to surgery, or oral Coumadin (warfarin) and/or Factor Xa inhibitors within 3 days prior to surgery.
3. Subject on antiplatelet/P2Y12 inhibitors medication 5 days prior to surgery;
4. Subject is currently participating or plans to participate in any other investigational product or drug trial without prior approval from the Sponsor.
5. Subjects who are known, current alcohol and/or drug abusers.
6. Subjects with any pre-operative findings identified by the surgeon that may preclude conduct of the study procedure.
7. Subjects with any intra-operative findings identified by the surgeon that may preclude the use of study product.
8. Subject with TBS in an actively infected field (Class III Contaminated or Class IV Dirty or Infected; see Appendix 1).
9. TBS is on arteries or veins where application of SURGICEL Powder would present a risk of introducing the study product into an open blood vessel.
10. Major arterial or venous bleeding or major defects in arteries and veins.
11. TBS where silver nitrate or any other escharotic chemicals have been applied.
12. TBS is in, around, or in proximity to foramina in bone, or areas of bony

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Drum Tower Hospital - Nanjing University Medical School, Nanjing
  - Ruijin Hospital - Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Xinhua Hospital, Shanghai
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened up to 21 days prior to surgery and attended a baseline visit within 24 hours of surgery. Both visits took place at a clinic within the hospital where surgery also took place. Subjects were followed until hospital discharge and requested to attend a visit at 30 (+14) days post surgery and at 6 months (+/- 30 days) either at the hospital or via telephone.
Pre-assignment Details: Subjects required to meet pre-defined inclusion/exclusion criteria prior to receiving study product. Subjects required to have an appropriate mild or moderate target bleeding site (TBS) identified intra-operatively. Subjects excluded if the TBS was where silver nitrate or any other escharotic chemicals were applied, was in, around, or in proximity to foramina in bone, areas of bony confine.
Groups:
- SURGICEL Powder: SURGICEL Powder Absorbable Hemostat (Oxidized Regenerated Cellulose)
- SURGICEL Original: Absorbable Hemostat (Oxidized Regenerated Cellulose)
Period: Overall Study
Arm/Group | SURGICEL Powder | SURGICEL Original
Started | 119 | 115
Completed (6 month follow-up) | 117 | 114
Not Completed | 2 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SURGICEL Powder | SURGICEL Original | Total
Number analyzed (Participants) | 119 | 115 | 234
Age, Continuous [Median (Full Range); unit: Years] | 54.0 [20 to 96] | 52.0 [23 to 89] | 53.0 [20 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 73 | 150
  Male | 42 | 42 | 84
Race/Ethnicity, Customized [Number; unit: Participants]
  Han | 116 | 114 | 230
  Other | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hemostatic Success at 5 Minutes
Description: Percentage of subjects achieving hemostatic success at 5 minutes following study product application with no rebleeding requiring additional treatment at the Target Bleeding Site (TBS) any time prior to initiation of final fascial closure
Time Frame: From product application to 5 minutes following product application
Population: Per Protocol Analysis (All intent to treat subjects who have no major protocol deviations and have data available for primary effectiveness endpoint)
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder | SURGICEL Original
Number analyzed (Participants) | 114 | 115
Participants | 109 | 103
Statistical Analysis 1: Comparison: SURGICEL Powder vs SURGICEL Original; Test type: Non-Inferiority — 10% margin; p < 0.0001, Farrington-Manning method — Testing whether the group difference in proportion of successes is >-0.1 (Test Group - Control Group); Risk Difference (RD) = 0.0605, 97.5% CI 1-sided [lower limit -0.0189]

2. Secondary Outcome: Hemostatic Success at 3 Minutes
Description: Percentage of subjects achieving hemostatic success at 3 minutes following study product application with no rebleeding requiring additional treatment at the TBS any time prior to initiation of final fascial closure
Time Frame: From product application to 3 minutes following product application
Population: Intent to Treat Analysis (All randomized and enrolled subjects for whom TBS was identified. Subjects who did not complete the procedure after TBS identification were included in the ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder | SURGICEL Original
Number analyzed (Participants) | 119 | 115
Participants | 107 | 92
Statistical Analysis 1: Comparison: SURGICEL Powder vs SURGICEL Original; Test type: Other; Farrington-Manning Method; Difference in proportion of successes (Test Group - Control Group); Difference in proportion of successes = 0.0992, 95.0% CI 2-sided [0.0078 to 0.1906]

3. Secondary Outcome: Hemostatic Success at 10 Minutes
Description: Percentage of subjects achieving hemostatic success at 10 minutes following study product application with no rebleeding requiring additional treatment at the TBS any time prior to initiation of final fascial closure
Time Frame: From product application to 10 minutes following product application
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder | SURGICEL Original
Number analyzed (Participants) | 119 | 115
Participants | 114 | 107
Statistical Analysis 1: Comparison: SURGICEL Powder vs SURGICEL Original; Test type: Other; Farrington-Manning Method; Difference in proportion of successes (Test Group - Control Group); Difference in proportion of successes = 0.0275, 95% CI 2-sided [-0.0312 to 0.0863]

4. Other Pre Specified Outcome: Number of Participants With Thromboembolic Events
Description: Number of participants with thrombotic events assessed as unlikely, possibly, probably or related to the study treatment
Time Frame: From enrollment to 30-day follow-up visit
Population: Safety Analysis Set (All enrolled subjects who underwent study procedure and received study product, and had post-baseline data. Enrollment defined as subjects with completed informed consent and meets all inclusion criteria and does not meet any exclusion criteria)
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder | SURGICEL Original
Number analyzed (Participants) | 119 | 115
Participants
  Investigator Assessment | 0 | 0
  Sponsor Assessment | 0 | 0

5. Other Pre Specified Outcome: Number of Participants With Post-operative Re-bleeding Events
Description: Number of participants with post-operative re-bleeding events assessed as unlikely, possibly, probably or related to study treatment and requiring medical/surgical intervention
Time Frame: From initiation of final fascial closure to 30-day follow-up visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder | SURGICEL Original
Number analyzed (Participants) | 119 | 115
Participants
  Investigator Assessment | 1 | 1
  Sponsor Assessment | 1 | 0

6. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events Requiring Surgical Intervention
Description: Number of Participants with Serious Adverse Events requiring surgical intervention and assessed as being unlikely, possibly, probably or related to study treatment
Time Frame: From enrollment to 6 month follow up visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder | SURGICEL Original
Number analyzed (Participants) | 119 | 115
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (serious and non-serious), whether attributable to device/procedure or not, were recorded from enrollment (informed consent and subject met all incl/excl criteria), during surgical procedure, and until completion of 30-day follow-up visit. Between 30 day and 6 month visit, all SAEs requiring surgical intervention and assessed as possibly/related to study treatment were recorded. All deaths were recorded regardless of relationship to product or procedure.
Description: For this study, an adverse event was any untoward medical occurrence (sign, symptom or disease) in a subject and which does not necessarily have a causal relationship with the study medical device. An untoward medical occurrence includes any new, undesirable medical experience or worsening of a pre-existing condition.
Arm/Group | SURGICEL Powder | SURGICEL Original
All-Cause Mortality (participants affected / at risk) | 2/119 | 1/115
Serious Adverse Events (participants affected / at risk) | 9/119 | 5/115
Other Adverse Events (participants affected / at risk) | 83/119 | 80/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURGICEL Powder (N=119) | SURGICEL Original (N=115)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhagic Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary Air Leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anastomotic Fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Shock Hemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Venous Thrombosis Limb (Vascular disorders) | 1 (1) | 0 (0)
Hemophilia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURGICEL Powder (N=119) | SURGICEL Original (N=115)
Incision Site Pain (Injury, poisoning and procedural complications) | 33 (34) | 26 (28)
Incision Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural Hypertension (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision Site Hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pancreatic Leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (8) | 6 (6)
Abdominal Distension (Gastrointestinal disorders) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 7 (9) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (4)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis Noninfective (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysbacteriosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Phase Reaction (General disorders) | 14 (14) | 12 (13)
Pyrexia (General disorders) | 7 (8) | 9 (9)
Asthenia (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (9) | 6 (7)
Hypoproteinaemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Metabolic Acidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 4 (4) | 8 (8)
Inflammatory Marker Increased (Investigations) | 4 (4) | 4 (4)
Blood Pressure Increased (Investigations) | 2 (2) | 3 (4)
Blood Potassium Decreased (Investigations) | 2 (2) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 1 (1)
C-reactive Protein Increased (Investigations) | 0 (0) | 1 (1)
Coagulation Test Abnormal (Investigations) | 0 (0) | 1 (1)
Protein Total Decreased (Investigations) | 1 (1) | 0 (0)
Urine Output Decreased (Investigations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 6 (6) | 1 (1)
Abdominal Infection (Infections and infestations) | 4 (4) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Fallopian Tube Abscess (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Reperfusion Injury (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Poor Quality Sleep (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Initial Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator and institution will not be able to publish single-center study data until combined results of the multicenter study are published. If multicenter publication is not performed within 12 months after the end or if sponsor notifies principal investigator and institution in writing that the multicenter study results will not be published, the principal investigator and institution may publish the results of their studies separately in accordance with contract.

DOCUMENTS (2):
  • Study Protocol (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT03783039/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03783039/SAP_001.pdf